A cover page

official title: Comparison of a SegNet-based Algorithm Estimating Epifascial Fibrosis

NCT number: NCT ID is pending, but not yet assigned.

document date: March 19th, 2021

Statistical Analysis Plan

Sample size was calculated using Power Analysis and Sample Size Software version 11.0.

(PASS, NCSS Statistical Software, Kaysville, UT, USA). As for two correlations analysis,

power of 0.80, α of 0.05, R0 (baseline correlation) of 0 and R1 (alternative correlation) of 0.5

were made, referred from the data of Koo et al.'s trial. The estimated lowest minimum sample

size is 29. Taken into consideration image processing-based trials are under easy control, mid-

term drop-out was expected to occur in very low chance. Allowing for a drop-out ratio of 5%,

30 patients were required. Two-sided statistical analyses were conducted using the Statistical

Package for the Social Sciences, version 24 (SPSS Inc., Chicago, USA). The normality

verification was performed using Kolmogorov-Smirnov. To remove linear effect derived from

interstitial fluid (BEI) or limb swelling (SCDR), the four types of index defined above were

compared to the BEI and SCDR using partial correlation analysis. If normal distribution was

not verified, they were analyzed after log transformation. A small positive number was added

before log transformation, if values were negative.